CLINICAL TRIAL: NCT07306234
Title: Efficacy and Safety of Doxycycline Versus Macrolides for Mycoplasma Pneumoniae Infection in Children (DOMINO): A Protocol for a Multicenter, Randomized, Open-Label, Superiority Trial
Brief Title: Doxycycline vs. Macrolide for MRMP (DOMINO)
Acronym: DOMINO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Young June Choe (Other)
Collaborators: Korea Society of Pediatric Infectious Diseases (Unknown); Korea National Institute of Health (Unknown); Korea Disease Control and Prevention Agency (Unknown); DT&CRO (Unknown)
Responsible Party: Sponsor-Investigator, Young June Choe, Professor, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOMINO; KNIH (Other Grant/Funding Number: National Institute of Health, Korea Disease Control and Prevention Agency)
Record Dates: First submitted 2025-12-22; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Mycoplasma Pneumoniae; Mycoplasma Pneumoniae Pneumonia
Keywords: Mycoplasma pneumoniae; Macrolide resistance; Children
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Doxycycline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Doxycycline) (Experimental): Participants will receive oral doxycycline (4 mg/kg/day divided into 2 doses for weight ≤45 kg; 100 mg BID for weight >45 kg). The standard treatment duration is 7 days, which may be extended up to 14 days based on clinical response.
  Interventions: Drug: Doxycycline
- Control Group (Azithromycin) (Active Comparator): Participants will receive oral azithromycin according to the standard 5-day regimen (10 mg/kg on Day 1, followed by 5 mg/kg on Days 2-5).
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Doxycycline — Intervention Group (Doxycycline): Participants will receive oral doxycycline (4 mg/kg/day divided into 2 doses for weight ≤45 kg; 100 mg BID for weight >45 kg). The standard treatment duration is 7 days, which may be extended up to 14 days based on clinical response.
  Arms: Intervention Group (Doxycycline)
Drug: Azithromycin — Control Group (Azithromycin): Participants will receive oral azithromycin according to the standard 5-day regimen (10 mg/kg on Day 1, followed by 5 mg/kg on Days 2-5).
  Rescue Therapy Protocol: To ensure patient safety, a standardized "rescue therapy" protocol is implemented. Participants in the Control group who fail to demonstrate clinical improvement at the 48-72 hour assessment-defined as persistent fever (≥38.0°C) or clinical deterioration-will be immediately switched to doxycycline. Consistent with the intention-to-treat principle, these cases will be classified as treatment failures for the primary efficacy analysis.
  Arms: Control Group (Azithromycin)

SUMMARY:
The goal of this clinical trial is to learn if doxycycline works to treat pneumonia in children. It focuses on children with Mycoplasma pneumoniae infection that may not respond to standard medicines. The main questions it aims to answer are:

* Does doxycycline stop fevers faster than azithromycin?
* Is doxycycline safe for children, specifically regarding tooth color changes?

Researchers will compare doxycycline to azithromycin to see if doxycycline works better to treat this type of pneumonia.

Participants will:

* Take either doxycycline or azithromycin by mouth for 7 to 14 days.
* Check their body temperature to see when their fever goes away.
* Visit the hospital to check for any medical problems.
* Have their teeth checked for color changes 28 days after starting the medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 to 17 years at the time of enrollment.
* Diagnosis: Clinically diagnosed CAP characterized by respiratory symptoms (e.g., fever, cough, auscultatory findings) and chest X-ray confirming pulmonary infiltrates.
* Pathogen: Confirmed MP M. pneumoniae infection via PCR OR strongly suspected infection based on clinical features and epidemiological grounds (e.g., outbreaks among classmates, poor response to prior non-macrolide antibiotics).
* Resistance: Suspected macrolide-resistant M. pneumoniae (MRMP) infection (e.g., during a reported local epidemic of MRMP).
* Timing: Ability to register and initiate the study drug within 72 hours of symptom onset.

Exclusion Criteria:

* Prior use of tetracyclines, macrolides, or quinolones for the current illness.
* Complicated pneumonia (e.g., necrosis, empyema, lung abscess) or severe pneumonia requiring immediate intensive care or exhibiting hypoxia (SpO₂ <90%).
* Hypersensitivity or contraindications to macrolides or tetracyclines.
* Severe immunocompromised state or severe underlying lung disease.
* Severe hepatic impairment (AST/ALT >3x upper limits) or severe renal impairment.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Defervescence rate | 72 hours
  Defervescence rate at 72 hours. Defervescence is defined as the maintenance of body temperature below 38.0°C for at least 24 consecutive hours without antipyretics.

SECONDARY OUTCOMES:
Hospitalization Rate | Up to 30 days
  Percentage of participants requiring hospitalization due to the progression of pneumonia or complications.
Length of Hospital Stay | Up to 30 days
  The duration of hospitalization from admission to discharge.
Hospital Readmission Rate | Up to 30 days
  Percentage of participants readmitted to the hospital after initial discharge due to worsening of pneumonia.
Treatment Failure Rate at Day 7 | 7 days
  Treatment failure is defined as the occurrence of any of the following: need for rescue therapy (switching to doxycycline for the control group), addition of other antibiotics or systemic steroids, or clinical deterioration requiring intensive care unit (ICU) admission.
Time to Resolution of Respiratory Symptoms | Up to 30 days
  Time to resolution of respiratory symptoms (cough, dyspnea) assessed using a 4-point Likert scale. Resolution is defined as the point at which the symptom score reaches 0 (none) or 1 (mild) and is maintained
Time to Radiological Resolution of Infiltrates | Up to 30 days
  Time to resolution of pulmonary infiltrates as confirmed by chest radiography follow-up.
Incidence of Tooth Discoloration in Children Under 8 Years | Day 28
  Assessment of visible tooth discoloration evaluated by visual inspection.

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Department of Pediatrics, Pusan National University School of Medicine, Pusan National University Children's Hospital, Yangsan, Republic of Korea, Busan
  - Department of Pediatrics, Gyeongsang National University College of Medicine, Gyeongsang National University Changwon Hospital, Changwon, Republic of Korea, Changwon
  - Department of Pediatrics, Chosun University College of Medicine, Chosun University Hospital, Gwangju, Republic of Korea, Gwangju
  - Department of Pediatrics, Jeju National University School of Medicine, Jeju National University Hospital, Jeju, Republic of Korea, Jeju City
  - Department of Pediatrics, CHA University School of Medicine, CHA Bundang Medical Center, Seongnam, Republic of Korea, Seongnam
  - Department of Pediatrics, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Republic of Korea, Seongnam
  - Department of Pediatrics, College of Medicine, The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Republic of Korea, Seoul
  - Department of Pediatrics, College of Medicine, The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Republic of Korea, Seoul
  - Department of Pediatrics, Eulji University School of Medicine, Eulji University Hospital, Seoul, Republic of Korea, Seoul
  - Department of Pediatrics, Korea University College of Medicine, Korea University Anam Hospital, Seoul, Republic of Korea, Seoul
  - Department of Pediatrics, Korea University College of Medicine, Korea University Guro Hospital, Seoul, Republic of Korea, Seoul
  - Department of Pediatrics, Seoul National University College of Medicine, Seoul National University Children's Hospital, Seoul, Republic of Korea, Seoul
  - Department of Pediatrics, Sungkyunkwan University School of Medicine, Samsung Medical Center, Seoul, Republic of Korea, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the publication will be made available to researchers who provide a methodologically sound proposal. This includes text, tables, figures, and appendices. IPD will be available beginning 6 months and ending 36 months following article publication.
  Supporting Information: The study protocol, statistical analysis plan (SAP), and informed consent form will also be shared. Access Criteria: Proposals should be directed to the Principal Investigator at [Insert Official Email Address]. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Wormser GP, Dattwyler RJ, Shapiro ED, Halperin JJ, Steere AC, Klempner MS, Krause PJ, Bakken JS, Strle F, Stanek G, Bockenstedt L, Fish D, Dumler JS, Nadelman RB. The clinical assessment, treatment, and prevention of lyme disease, human granulocytic anaplasmosis, and babesiosis: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2006 Nov 1;43(9):1089-134. doi: 10.1086/508667. Epub 2006 Oct 2. PMID 17029130
- [Result] Cummings MM. Copyright and reproduction. Bull Med Libr Assoc. 1973 Jul;61(3):344-5. No abstract available. PMID 4725345
- [Result] Kang DH, Lee JY, Chung JH, Cho JM, Lee SH, Park J, Kim TH, Yoo TK, Lee SW. Comparison of efficacy for erectile function and lower urinary tract symptoms of tadalafil 20 mg on-demand and 5 mg once daily in patients with erectile dysfunction. Int J Clin Pract. 2012 Aug;66(8):813-820. doi: 10.1111/j.1742-1241.2012.02946.x. PMID 22805273
- [Result] Xue H, Xu H, Song X, Chen M, Wang X, Ji M, Wang M. Porous Frustrated Lewis Pairs Catalyst Constructed on Defective Zirconium-Based Metal-Organic Frameworks for Hydrogenation Reactions with H2. Inorg Chem. 2024 Aug 26;63(34):16011-16017. doi: 10.1021/acs.inorgchem.4c02470. Epub 2024 Aug 15. PMID 39145892
- [Result] Guo T, Zamuner F, Ting S, Chen L, Rooper L, Tamayo P, Fakhry C, Gaykalova D, Mehra R. Clinical and genomic characterization of chemoradiation-resistant HPV-positive oropharyngeal squamous cell carcinoma. Front Oncol. 2024 Mar 5;14:1336577. doi: 10.3389/fonc.2024.1336577. eCollection 2024. PMID 38505587
- [Result] Forde E, Humphreys H, Greene CM, Fitzgerald-Hughes D, Devocelle M. Potential of host defense peptide prodrugs as neutrophil elastase-dependent anti-infective agents for cystic fibrosis. Antimicrob Agents Chemother. 2014;58(2):978-85. doi: 10.1128/AAC.01167-13. Epub 2013 Nov 25. PMID 24277028
- [Result] Liu Y. [Lay further emphasis on the cosmetic repair of deep burn wounds in extraordinary regions or caused by uncommon agents]. Zhonghua Shao Shang Za Zhi. 2014 Oct;30(5):389-91. Chinese. PMID 25572886
- [Result] Jiao R, Xue B, Zhang M. A Multiform Optimization Framework for Constrained Multiobjective Optimization. IEEE Trans Cybern. 2023 Aug;53(8):5165-5177. doi: 10.1109/TCYB.2022.3178132. Epub 2023 Jul 18. PMID 35687640
- [Result] Han S, Luo Y, Liu B, Guo T, Qin D, Luo F. Dietary flavonoids prevent diabetes through epigenetic regulation: advance and challenge. Crit Rev Food Sci Nutr. 2023 Nov;63(33):11925-11941. doi: 10.1080/10408398.2022.2097637. Epub 2022 Jul 11. PMID 35816298
- [Result] Morozumi M, Hasegawa K, Kobayashi R, Inoue N, Iwata S, Kuroki H, Kawamura N, Nakayama E, Tajima T, Shimizu K, Ubukata K. Emergence of macrolide-resistant Mycoplasma pneumoniae with a 23S rRNA gene mutation. Antimicrob Agents Chemother. 2005 Jun;49(6):2302-6. doi: 10.1128/AAC.49.6.2302-2306.2005. PMID 15917525
- [Result] Tolbert K, Stubbs E. Rational use of gastroprotectants in cats: An evidence-based approach. J Feline Med Surg. 2024 Aug;26(8):1098612X241274235. doi: 10.1177/1098612X241274235. PMID 39105658
- [Result] MacGowan AP, Noel AR, Tomaselli S, Bowker KE. Pharmacodynamics of ceftaroline against Staphylococcus aureus studied in an in vitro pharmacokinetic model of infection. Antimicrob Agents Chemother. 2013 Jun;57(6):2451-6. doi: 10.1128/AAC.01386-12. Epub 2013 Mar 4. PMID 23459495
- [Result] Roddy SP, Darling RC 3rd, Chang BB, Kreienberg PB, Paty PS, Lloyd WE, Shah DM. Brachial artery reconstruction for occlusive disease: a 12-year experience. J Vasc Surg. 2001 Apr;33(4):802-5. doi: 10.1067/mva.2001.112705. PMID 11296335